CLINICAL TRIAL: NCT03643562
Title: Open-label Evaluation of Adrabetadex in Patients With Neurologic Manifestations of Niemann-Pick Type C Disease (NPC)
Brief Title: Niemann-Pick Type C Treatment With Adrabetadex for Symptoms of Brain and Nervous System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor had determined that the benefit-risk profile of adrabetadex was not favorable and the clinical development program for adrabetadex was discontinued.
Sponsor: Mandos LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTS-270-001
Record Dates: First submitted 2018-08-19; First posted 2018-08-23 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Niemann-Pick Type C Disease
Keywords: Niemann-Pick; NPC; NPC Type 1 (NPC1)
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Intervention Model Description: Continued treatment for children at least 4 years of age
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adrabetadex (Experimental): Participants will receive prescribed adrabetadex by intra-thecal (IT) injection every 2 weeks.
  Interventions: Drug: Adrabetadex

INTERVENTIONS:
Drug: Adrabetadex — Administered via lumbar puncture (LP) and IT infusion
  Other Names: VTS-270

SUMMARY:
This study was amended from expanded access to a clinical trial. Information will be collected about long-term safety and effectiveness of adrabetadex shots in the spine every 2 weeks.

Participants who were already taking adrabetadex will receive their stable dose. Participants who have not ever taken it will start by receiving 400 mg.

Participants will receive treatment every 2 weeks until their doctor finds it does not help them anymore, they withdraw, or the study is stopped for any reason. Participants will not receive additional study treatment after their participation in this protocol.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, a participant must meet the following criteria:

* Is male or female and at least 4 years of age at time of screening.
* Has a confirmed diagnosis of NPC and exhibits neurologic symptoms.
* Has written informed consent/assent to participate.
* Has the ability to undergo LP and IT drug administration.
* If taking miglustat (Zavesca®), must have been on a stable dose for the past 6 weeks and be willing to remain on a stable dose for the duration of participation in the study, or discontinue miglustat use at least 6 weeks before entry into the study (Day 1).
* If has a history of seizures, the condition is adequately controlled as per protocol requirements.
* Agrees to discontinue any investigational treatments (other than adrabetadex) for at least 1 month before first dose on Day 1.
* If engaging in heterosexual sex, agrees to use a protocol-defined method of contraception throughout the study, and until 30 days after completing the study.
* Has a responsible adult who the investigator determines is able and willing to comply with study requirements and a parent/guardian who will accompany the participant to study visits.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

* Weighs less than 15 kg.
* Has a history of hypersensitivity reactions to any product containing 2-hydroxypropyl-β-cyclodextrin (HP-β-CD) or has a history of hypersensitivity reactions or allergy to anesthesia/sedation.
* Has received treatment with any investigational product (other than adrabetadex) within 1 month prior to Day 1 of treatment.
* Is pregnant or nursing.
* Has systemic infection or uncontrolled psychosis.
* Has known history of a bleeding disorder.
* Has used anticoagulants within 2 months of entry into the study.
* Per protocol, or in the opinion of the investigator:

  1. has laboratory values that would preclude participation
  2. has suspected infection of the central nervous system (CNS)
  3. has a spinal deformity that could impact performance of repeated LPs
  4. has a serious skin infection in the lumbar region or evidence of obstructive or normal pressure hydrocephalus
  5. is unable to comply with the study requirements
  6. has a medical condition that might increase the risk of participation

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Mandos LLC
Locations (17):
- United States (17):
  - University of Arkansas System, Little Rock, Arkansas
  - Loma Linda University Health System, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Children's Specialty Center of Nevada, Las Vegas, Nevada
  - NYU Langone Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Carilion Medical Center, Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Naive: Treatment-naive participants received prescribed adrabetadex by intra-thecal (IT) injection via lumbar puncture (LP) every 2 weeks. Treatment with adrabetadex continued until the clinician considered adrabetadex to be no longer beneficial to the participant, the participant withdrew from the study, adrabetadex received marketing authorization in the United States, or the development program was discontinued.
- Previously Treated: Previously-treated participants received prescribed adrabetadex by IT injection via LP every 2 weeks. Treatment with adrabetadex continued until the clinician considered adrabetadex to be no longer beneficial to the participant, the participant withdrew from the study, adrabetadex received marketing authorization in the United States, or the development program was discontinued.
Period: Overall Study
Arm/Group | Treatment Naive | Previously Treated
Started | 9 | 18
Received at Least 1 Dose of Study Drug | 9 | 18
Completed | 1 | 2
Not Completed | 8 | 16
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Study Terminated by Sponsor | 2 | 10
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other than specified | 3 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Treatment Naive: Treatment-naive participants received prescribed adrabetadex by IT injection via LP every 2 weeks. Treatment with adrabetadex continued until the clinician considered adrabetadex to be no longer beneficial to the participant, the participant withdrew from the study, adrabetadex received marketing authorization in the United States, or the development program was discontinued.
- Total: Total of all reporting groups
Arm/Group | Treatment Naive | Previously Treated | Total
Number analyzed (Participants) | 9 | 18 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.33 (8.718) | 17.94 (13.705) | 16.07 (12.388)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 18 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 17 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as an AE with onset on or after the start of adrabetadex treatment. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 134
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Naive | Previously Treated
Number analyzed (Participants) | 9 | 18
Participants
  All TEAEs | 9 | 17
  SAEs | 5 | 9

ADVERSE EVENTS:
Time Frame: Baseline up to Week 134
Description: All enrolled participants
Arm/Group | Treatment Naive | Previously Treated
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/18
Serious Adverse Events (participants affected / at risk) | 5/9 | 9/18
Other Adverse Events (participants affected / at risk) | 9/9 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (N=9) | Previously Treated (N=18)
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Norovirus test positive (Investigations) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Lennox-Gastaut syndrome (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 3
Mental status changes (Psychiatric disorders) | 0 | 1
Staring (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (N=9) | Previously Treated (N=18)
Tachycardia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 2
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 2 | 4
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Gaze palsy (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 4
Adverse drug reaction (General disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 7
Gait disturbance (General disorders) | 1 | 1
Gait inability (General disorders) | 0 | 1
Medical device site injury (General disorders) | 1 | 0
Procedural failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Unevaluable event (General disorders) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 8
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1
Intentional product use issue (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Coronavirus test positive (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 5 | 6
Balance disorder (Nervous system disorders) | 0 | 1
Cataplexy (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Hypersomnia (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Primary headache associated with sexual activity (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Communication disorder (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne cystic (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This study was terminated early when the Sponsor had determined that the benefit-risk profile of adrabetadex was not favorable and the clinical development program for adrabetadex was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03643562/Prot_SAP_001.pdf